CLINICAL TRIAL: NCT02466906
Title: Recombinant Human Granulocyte-macrophage Colony-stimulating Factor as Adjuvant Immunotherapy in Treating Resectable Stage III Colon Cancer: A Randomized, Placebo-controlled Clinical Trial
Brief Title: RhGM-CSF as Adjuvant Immunotherapy in Treating Stage III Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L-15-01
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Colon Cancer
Keywords: Stage III colon cancer; rhGM-CSF; Immunotherapy; Surgery; Adjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — regramostim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhGM-CSF group (Experimental): rhGM-CSF was injected subcutaneously perioperation.
  Interventions: Drug: rhGM-CSF
- placebo group (Placebo Comparator): Placebo was injected subcutaneously perioperation.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhGM-CSF — rhGM-CSF was injected subcutaneously of 3± 0.3ug/kg/d per day for 5 days before and 2 days after surgery. During adjuvant therapy of XELOX, rhGM-CSF was continuous injected for 6 days when finishing each cycle of chemotherapy (from d15) or stopped when ANC>20.0X109/L.
  Arms: rhGM-CSF group
Drug: placebo — Placebo was injected subcutaneously of 3± 0.3ug/kg/d per day for 5 days before and 2 days after surgery. . During adjuvant therapy of XELOX, placebo was continuous injected for 6 days when finishing each cycle of chemotherapy (from d15).
  Arms: placebo group

SUMMARY:
This study is to investigate the efficacy and safety of rhGM-CSF as adjuvant immunotherapy for patients with resectable stage III colon cancers.

DETAILED DESCRIPTION:
This study is to investigate the efficacy and safety of rhGM-CSF as adjuvant immunotherapy for patients with resectable stage III colon cancers. Patients were randomly assigned to rhGM-CSF group or placebo group and treated with rhGM-CSF or placebo perioperation and during the adjuvant chemotherapy. The purpose of the study is to evaluate the antitumor immune effect of rhGM-CSF before surgery and adjuvant chemotherapy through DFS of 5 years and to observe the safety during the treatment in order to provide evidence for improvement in treating resectable colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as resectable stage III colon cancer
2. 18-70 years old
3. ECOG performance status ≤2
4. Unexposed to rhGM-CSF in 6 months
5. Signed an informed consent document

Exclusion Criteria:

1. Secondary primary cancer, or concurrent primary malignancies (except for basal cell or squamous cell skin cancer, cervical cancer in situ, and other cancer with disease free for more than 5 years)
2. Complete intestinal obstruction
3. Events within 6 months before randomization: myocardial infarction, sever or unstable angina, coronary artery or peripheral arterial bypass surgery, congestive heart failure ( NYHA functional class of III or IV ), stroke and any myocardial dysfunction in a transient ischaemic attack
4. Abnormal liver and kidney function (Serum creatinine > 1.5 x ULN, total bilirubin > 1.5 x ULN, transaminase > 3 x ULN ), abnormal pulmonary function (FEV1<60% or diffusing capacity of the lung for carbon monoxide < 55% )
5. Bone marrow dysfunction ( Hb<9.0 g/dL、ANC<1.5 x 109/L、PLT<100 x 109/L )
6. ITP or immunodeficiency
7. Uncontrolled infection, including HBV, HCV, HIV infection
8. Female patients who has been pregnant or planning to, and those during lactation
9. Known allergic to E.coli agents or rhGM-CSF or any severe allergic history to other drugs
10. Other cases that the researcher found ineligible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival（DFS） | 5 years

SECONDARY OUTCOMES:
Immune anti-tumor effect: DC cells, CD4+ cells, CD8+ cells, Treg cells | 5
Overall survival (OS) | 5 years
Incidence of liver metastasis | 5 years
Adverse effects (AE) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China